CLINICAL TRIAL: NCT04119947
Title: Evaluation of Safety, Tolerance and Pharmacokinetics/Pharmacodynamics of SY-009 Capsules After Single Dose Incremental Oral Administration in Healthy Subjects
Brief Title: Single Ascending Oral Doses of SY-009 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Yabao Pharmaceutical R&D Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SY009001
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2018-11

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Parallel ，Placebo control
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- SY-009 dose 1 (Experimental): A single dose of SY-009 (0.5-40mg) taken orally.
  Interventions: Drug: SY-009
- SY-009 dose 2 (Experimental): A single dose of SY-009 (0.5-40mg) taken orally.
  Interventions: Drug: SY-009
- SY-009 dose 3 (Experimental): A single dose of SY-009 (0.5-40mg) taken orally.
  Interventions: Drug: SY-009
- SY-009 dose 4 (Experimental): A single dose of SY-009 (0.5-40mg) taken orally.
  Interventions: Drug: SY-009
- SY-009 dose 5 (Experimental): A single dose of SY-009 (0.5-40mg) taken orally.
  Interventions: Drug: SY-009
- SY-009 dose 6 (Experimental): A single dose of SY-009 (0.5-40mg) taken orally.
  Interventions: Drug: SY-009
- SY-009 matching placebo (Placebo Comparator): from 2-40mg
  Interventions: Drug: SY-009

INTERVENTIONS:
Drug: SY-009 — The study will be initiated in healthy subjects at a 0.5mg dose that is the maximum recommended starting dose(MRSD) . Doses will be escalated in subsequent dosing process, after appropriate review of safety data. The subsequent planned doses are 2,5, 10, 20, 40mg successively. The increment of the dose escalation may be reduced, a lower dose may be administered following data review.

SUMMARY:
This is a phase Ⅰ，single-center, randomized, double-blinded, placebo-controlled, single ascending dose trial of SY-009 in healthy subjects.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, dosed tolerability, pharmacokinetic / pharmacodynamic study of a single oral SY-009 capsule for Chinese healthy subjects. Plan to screening no more than 64 healthy subjects ， dividing them into 7 dose groups.

ELIGIBILITY:
Inclusion Criteria:

1、healthy subject：determined by medical history, physical examination, Imaging examination, abdominal B-mode ultrasonography (include liver, gallbladder, pancreas, spleen and kidney), electrocardiogram and laboratory tests. Test results within the normal range for the population or investigator site, or with abnormalities deemed clinically insignificant by the investigator; 2、Gender: Male and female, gender balance; 3、Age: 18-65 years old (including the boundary values); 4、Weight ≥50kg and 19.0kg/m2≤BMI≤28.0kg/m2 [BMI=body weight（kg）/height 2 (m2); 5、fasting plasm glucose (FPG): 3.9-6.1mmol/L (excluding the boundary valuses); 6、2h postprandial plasma giucose（2hPPG）<7.8mmol/L; 7、glycosylated hemoglobin (HbA1c) <5.7%;

8、have venous access sufficient to allow blood sampling as per the protocol;

9、Subjects must have informed consent before the study and sign a written informed consent form voluntarily;

10、Subjects can communicate well with investigator and complete the study according to the protocol.

Exclusion Criteria:

1. are investigator site personnel directly affiliated with this study and their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted.
2. within 3 months prior to screening, complete or withdraw a clinical study, or are currently conducting a clinical study. Or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
3. have previously completed or withdrawn from this study.
4. have known allergies to compounds related to SY-009 capsules or its adjuvants,or allergic constitution/allergic history, or SGLT1 or SGLT2 inhibitors taken in the past one year.
5. with cardiovascular diseases, respiratory diseases, gastrointestinal diseases, endocrine diseases, blood system diseases, nervous system diseases, disease status can significantly change the absorption, distribution, metabolism and excretion of experimental drugs, or taking experimental drugs will increase the risk of subjects.
6. In the past five years, there has been a history of drug abuse or drug abuse tests positive.
7. show evidence or test positive on any of the following: hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibody (HCV), Treponema pallidum antibody (S-TP), HIV (HIV1 + 2) antibody.
8. Blood donation or massive blood loss exceeding 400 mL in the first three months prior to screening, or surgical operation and blood or blood component transfusion within the first four weeks prior to screening, or have history of fainting or needle fainting.
9. Subjects who have an average weekly alcohol intake that exceeds and 14 units per week (1 unit = 360 mL beer, 45 mL alcohol content of 40% spirits or 150 mL wine) or subjects unwilling to stop alcohol consumption 24 hours prior to dosing until the completion of each inpatient study period.
10. consume more than 5 cigarettes per day or the equivalent, or are unable or unwilling to refrain from nicotine during the study.
11. intend to use any medicine or health care product within 14 days prior to dosing or during the study.
12. subjects not agree to use reliable contraceptive methods (hormones or barriers or abstinence) during the study period and at least 1 month after administration.
13. women were positive for blood pregnancy test within 24 hours prior to enrollment.
14. pregnant or lactating women.
15. Have special dietary requirements，and impossible to comply with the unified diet.
16. Unable to stop eating chocolate, any caffeine-containing food or beverage (such as pitaya, grapefruit, orange juice, mango, etc.) 48 hours before administration and during the study.
17. Within 30 days prior to screening, any drugs that inhibit or induce drug metabolic enzymes in the liver (e.g. barbiturates, carbamazepine, phenytoin sodium, glucocorticoids, omeprazole, SSRI antidepressants, cimetidine, diltiazem, macrolides, nitroimidazoles, sedative hypnotics, verapamil, fluoroquinolones, antihistamines) were used.
18. in the opinion of the investigator , are unsuitable for inclusion in the study，or subjects withdraw informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
The Safety and tolerance of SY-009，Collecting Number of subjects with adverse events as assessed by CTCAE V5.0 | 7 Days
  Number of subjects with adverse events, major adverse events, serious adverse events, pregnancy events, abnormal Laboratory Values, abnormal vital signs, Abnormal physical examination, Abnormal ECG data.

SECONDARY OUTCOMES:
area under curve (AUC) of SY-009 following oral administration of single ascending dose | 3 Days
  to measure the study drug concentration in blood samples to be collected after drug administration.
Cmax of SY-009 following oral administration of single ascending dose | 3 Days
  to measure the study drug concentration in blood samples to be collected after drug administration.
T1/2 of SY-009 following oral administration of single ascending dose | 3 Days
  to measure the study drug concentration in blood samples to be collected after drug administration.
CL/F (Clearance rectified) of SY-009 following oral administration of single ascending dose | 3 Days
  to measure the study drug concentration in blood samples to be collected after drug administration.
glucose levels following single dose of SY-009 | 3 Days
  FPG AUC
insulin secretion following single dose of SY-009 | 3 Days
  insulin changes
C-peptide secretion following single dose of SY-009 | 3 Days
  C-peptide change

CONTACTS AND LOCATIONS:
Overall Officials: Jingtong Li, Doctor, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China